CLINICAL TRIAL: NCT03520712
Title: A Phase 1/2 Safety, Tolerability, and Efficacy Study of Valoctocogene Roxaparvovec, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A Patients With Residual FVIII Levels ≤ 1 IU/dL and Pre-existing Antibodies Against AAV5
Brief Title: Gene Therapy Study in Severe Hemophilia A Patients With Antibodies Against AAV5
Acronym: GENEr8-AAV5+
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early rollover into long-term extension study
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270-203; 2017-000662-29 (EudraCT Number)
Record Dates: First submitted 2018-04-10; First posted 2018-05-11 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A; Gene Therapy; Clotting Disorders; Blood Disorder
Keywords: Hemophilia A; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn; Factor VIII; Coagulants; AAV5 antibodies
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders, Inherited; Blood Coagulation Disorders; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- valoctocogene roxaparvovec Open Label (Experimental): Single administration of BMN270 at a dose of 6E13 vg/kg
  Interventions: Biological: Valoctocogene Roxaparvovec

INTERVENTIONS:
Biological: Valoctocogene Roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
  Other Names: BMN 270

SUMMARY:
This study is being conducted by BioMarin Pharmaceutical Inc. as an open label, single dose study to determine the safety of valoctocogene roxaparvovec (an Adenovirus-Associated Virus (AAV) based gene therapy vector) in severe Hemophilia A patients with pre-existing antibodies against AAV5.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age with hemophilia A and residual FVIII levels ≤ 1 IU/dL as evidenced by medical history, at the time of signing the informed consent.
2. Detectable pre-existing antibodies against the AAV5 vector capsid as measured by AAV5 total antibody ELISA.
3. Subject must have been on prophylactic FVIII replacement therapy for at least 12 months prior to study entry.
4. No previous documented history of a detectable FVIII inhibitor, and results from a Bethesda assay or Bethesda assay with Nijmegen modification of less than 0.6 Bethesda Units (BU) (or less than 1.0 BU for laboratories with a historical lower sensitivity cutoff for inhibitor detection of 1.0 BU) on 2 consecutive occasions at least one week apart within the past 12 months (at least one of which should be tested at the central laboratory).
5. Sexually active participants must agree to use an acceptable method of effective contraception. Participants must agree to contraception use for at least 12 weeks post-infusion.

Exclusion Criteria:

1. Any evidence of active infection including COVID-19, or any immunosuppressive disorder, except for HIV infection. HIV positive patients who meet all other eligibility criteria may be included if they have a CD4 count > 200/mm3 and an undetectable viral load (unquantifiable viral load as defined as less than the limit of quantification by the testing laboratory's assay is permitted) while receiving an antiretroviral therapy (ART) regimen that does not contain efavirenz or another potentially hepatotoxic ART.
2. Evidence of liver dysfunction as assessed by liver tests and most recent, prior FibroScan or liver biopsy showing significant fibrosis of 3 or 4 as rated on a scale of 0-4 on the Batts-Ludwig (Batts 1995) or METAVIR (Bedossa 1996) scoring systems, or an equivalent grade of fibrosis if an alternative scale is used.
3. Chronic or active hepatitis B or C as evidenced by testing at screening.
4. Active malignancy, except non-melanoma skin cancer, or history of hepatic malignancy.
5. Any condition that, in the opinion of the investigator or Sponsor would prevent the patient from fully complying with the requirements of the study (including corticosteroid treatment and/or use of alternative immunosuppressive agents outlined in the protocol) and/or would impact or interfere with evaluation and interpretation of subject safety or efficacy result.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males only.
Enrollment: 3 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (9):
- Charlotte Maxeke Johannesburg Academic Hospital, Hemophilia Comprehensive Care Center, Johannesburg, South Africa
- South Korea (2):
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (2):
  - Royal Free Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 2 principal investigators at 2 study centers in 2 countries (South Africa and United Kingdom).
  Nine investigational sites were activated, 2 subjects in South Africa and 1 subject in the United Kingdom were enrolled in the study.
Pre-assignment Details: 10 participants were planned to be enrolled. 3 participants met all eligibility criteria & were enrolled in study. There were 26 screen failures.
Groups:
- BMN 270 6E13 vg/kg: BMN 270 6E13 vg/kg, given as a single intravenous dose (IV)
  Valoctocogene Roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
Period: Overall Study
Arm/Group | BMN 270 6E13 vg/kg
Started | 3
Completed | 1
Not Completed | 2
Not completed — Early termination of the study by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population was comprised of all participants who have received the BMN 270 infusion.
Arm/Group | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 2
  Black or African American | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1
  South Africa | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: A treatment-emergent adverse event (TEAE) is defined as any AE that newly appeared or worsened in severity following initiation of investigational product administration.
Time Frame: Up to 5 years post-infusion.
Population: The safety analysis was based on the ITT population.
  The intention-to-treat (ITT) population was comprised of all participants who have received the BMN 270 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 3
Participants
  Participants with any AE | 3
  Participants with any SAE | 1
  Participants with any treatment-related AE | 3
  Treatment-related SAEs | 1
  Participants with any AE of Grade >= 3 | 1
  AEs leading to dose adjustment during infusion | 0
  AEs leading to dose interruption during infusion | 0
  AEs leading to study drug discontinuation | 0
  Participants who died | 0

2. Secondary Outcome: Number of Participant With FVIII Activity >= 5 IU/dL at Week 26. Using Chromogenic Substrate Assay (CSA).
Description: Prior to BMN270 infusion, screening FVIII activity levels where participants had not received exogenous FVIII within 72 hours of assessment were below the lower limit of quantitation (LLOQ) as measured by CSA (LLOQ = 0.015 IU/mL).
Time Frame: 26 weeks
Population: The intention-to-treat (ITT) population was comprised of all participants who have received the BMN 270 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 3
Participants
  Participant with FVIII activity >= 5 IU/dL | 1
  Participant with FVIII activity < 5 IU/dL | 2

3. Secondary Outcome: Mean Annualized Factor VIII Utilization During Week 5 and Beyond
Description: The annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy is defined as Sum of FVIII use (IU/kg) during calculation period/Total number of days during the calculation period ×365.25
Time Frame: Week 5 and Beyond (Follow-Up, up to 1782 Days)
Population: The intention-to-treat (ITT) population was comprised of all participants who have received the BMN 270 infusion.
Measure: Mean (Standard Deviation); unit: IU/kg/yr
Arm/Group | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 3
IU/kg/yr | 661.1 (912.92)

4. Secondary Outcome: Mean Annualized Factor VIII Infusion Rate During Week 5 and Beyond
Description: Annualized FVIII replacement infusion rate=(number of FVFIII replacement infusions during calculation period/sum(follow-up days) of the period)*365.25
Time Frame: Week 5 and Beyond (Follow-Up, up to 1782 Days)
Population: The intention-to-treat (ITT) population was comprised of all participants who have received the BMN 270 infusion.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 3
ml/min | 21.9 (30.61)

5. Secondary Outcome: Number of Participants Showed Reduction in the ABR Post-BMN 270 Infusion. Impact of BMN 270 on the Number of Bleeding Episodes Requiring Exogenous FVIII Therapy.
Description: Annualized bleeding rate (ABR) (counts/yr.)=Number of bleeding episodes during calculation period/Total number of days during the calculation period ×365.25
Time Frame: Week 5 and Beyond (Follow-Up, up to 1782 Days)
Population: The intention-to-treat (ITT) population was comprised of all participants who have received the BMN 270 infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 270 6E13 vg/kg
Number analyzed (Participants) | 3
Participants
  Participants showed reduction in the ABR post-BMN 270 infusion | 3
  Participants who did not show reduction in the ABR post-BMN 270 infusion | 0

ADVERSE EVENTS:
Time Frame: up to 5 years post-infusion.
Description: The safety analysis was based on the ITT population.
  A treatment-emergent adverse event (TEAE) is defined as any AE that newly appeared or worsened in severity following initiation of investigational product administration.
Arm/Group | BMN 270 6E13 vg/kg
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 6E13 vg/kg (N=3)
Hypersensitivity (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 6E13 vg/kg (N=3)
Alanine aminotransferase increased (Investigations) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Hernia (General disorders) | 1 (1)
Thermal burns (Injury, poisoning and procedural complications) | 1 (1)
Influenza (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
In accordance with the study enrollment stopping criteria in the 270-203 study protocol and the Data Monitoring Committee (DMC) recommendation, decided to terminate 270-203, since 2 of the 3 participants in Cohort 1 (AAV5 TAb≤500) had FVIII activity 5IU/dL after a minimum of 6 weeks post-BMN 270 infusion. The last participant visit, and 270-203 termination, occurred on 07 August 2024.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT03520712/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT03520712/SAP_001.pdf